CLINICAL TRIAL: NCT01913743
Title: The Effects of Mindsets on the Brain's Response to Food Cues
Acronym: MINDSETS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Principal Investigator, Kathryn E. Demos, Assistant Professor (Research), The Miriam Hospital
Other Study IDs: MINDSETS - TOS
Record Dates: First submitted 2013-07-25; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Obesity
Keywords: fMRI; cognitive strategies; obesity; weight loss; mindsets
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MINDSETS: overweight/obese

SUMMARY:
Previous studies have shown that obese individuals exhibit greater reward-related brain activity in response to food cues than lean individuals and our group has shown that successful weight loss maintainers who were previously obese and now maintain a healthy weight have increased control-related activity when viewing food cues. These findings suggest key roles for both reward-related brain areas and inhibitory control regions in eating behavior. However, no studies to date have examined (a) whether the response to food cues (i.e., cue-reactivity) can be changed in obese individuals, (b) which strategies are most effective at altering brain response to food cues, or (c) the neural mechanisms that support such change.

Given the omnipresent environmental cues to eat and the association between heightened reward-responsivity and obesity, it is critical to investigate ways to potentially alter food cue-reactivity in the obese. The most widely employed approach for behavioral weight loss treatment is Cognitive Behavioral Therapy (CBT), which incorporates strategies to control and change cognitions (e.g., avoid desire to eat tempting foods by focusing on something else). This approach is sometimes described as "change- focused" because modifying negative thoughts is assumed to thereby change associated maladaptive emotions and behaviors. Alternatively, emerging evidence suggests Acceptance and Commitment Therapy (ACT), which teaches participants to recognize and accept their cravings as feelings that need not be acted upon, may also be effective in treating obesity. A third strategy often employed in smoking cessation and substance abuse treatment is to focus on the long-term consequences of behaviors, however this form of treatment is not typically used in behavioral weight loss therapy. Thus although each approach is potentially effective, these treatment approaches differ greatly in the cognitive strategies they employ.

The primary aim of the proposed research is to compare a cognitive strategy used in CBT ('CHANGE'), a cognitive strategy emphasized in ACT ('ACCEPT'), and a cognitive strategy used in smoking cessation ('LATER') relative to a control condition ('NOW'), in their effectiveness in altering reward and inhibitory control responses to food cues among obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* MRI compatibility
* 25-55 yrs old
* 25-40 BMI
* weight stable
* right handed

Exclusion Criteria:

* MRI incompatibility
* left handed

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The recruited sample will include both males and females between the ages of 25-55 years with BMIs between 25-40. This age range reflects the modal ages for obese participants presenting for behavioral weight loss, and individuals with BMIs greater than 40 typically do not fit comfortably within the scanner bore. As with previous studies at the WCDRC, all participants will be weight stable (defined as within +/- 5 lbs. for the past two months).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) signal differences between 4 different mindset conditions in response to food cues | 1 day (single time point)
  brain response to food cues measured via functional magnetic resonance imaging (fMRI) BOLD signal change will be assessed across all participants while using the 4 different mindsets potential differences in the BOLD response to food cues will be assessed between the 4 mindsets

SECONDARY OUTCOMES:
behavioral measures of physical activity and eating behavior assessed via questionnaires | 1 day (single time point)
  behavioral measures of physical activity and eating behavior will be assessed via questionnaires in order to describe the sample

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn E Demos, PhD, Principal Investigator — Brown University Medical School
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States